CLINICAL TRIAL: NCT03354143
Title: Hypertension, Intracranial Pulsatility and Brain Amyloid-beta Accumulation in Older Adults (HIPAC Trial)
Acronym: HIPAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Texas Health Resources (Other); Michigan State University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Rong Zhang, Professor of Neurology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STU 102017-029; 5R01AG057571-05 (NIH)
Record Dates: First submitted 2017-11-15; First posted 2017-11-27 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Hypertension
Keywords: Dementia; Alzheimer's Disease; Blood Pressure; Cognitive Function; Magnetic Resonance Imaging
MeSH Terms: conditions — Hypertension; Dementia; Alzheimer Disease | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Care (Active Comparator): Subjects in the standard care arm will receive calcium channel blocker (CCB, amlodipine), angiotensin II receptor blocker (ARB, losartan), and other antihypertensive drugs to reduce 24-hour SBP ≤ 130 mmHg. Drug doses will be titrated to reach the BP target.
  Interventions: Other: Standard Care
- Intensive Treatment (Experimental): Subjects in the intensive treatment arm will receive calcium channel blocker (CCB, amlodipine), angiotensin II receptor blocker (ARB, losartan), and other antihypertensive drugs to reduce 24-hour SBP ≤ 120 mmHg.
  Interventions: Other: Intensive Treatment
- Control group subjects (No Intervention): Healthy normotensive subjects (24-hour ambulatory BP<125/75 mmHg without use of antihypertensive medication) who undergo MRI as part of standard of care.

INTERVENTIONS:
Other: Standard Care — Calcium channel blocker (CCB, amlodipine), angiotensin II receptor blocker (ARB, losartan), and other antihypertensive drugs will be used to reduce 24-hour SBP ≤ 130 mmHg.
  Arms: Standard Care
Other: Intensive Treatment — Calcium channel blocker (CCB, amlodipine), angiotensin II receptor blocker (ARB, losartan), and other antihypertensive drugs will be used to reduce 24-hour SBP ≤ 120 mmHg.
  Arms: Intensive Treatment

SUMMARY:
The aim of this study is to determine if lowering blood pressure using FDA approved medication (antihypertensive drugs) alters brain pulsatility and reduces brain amyloid beta protein accumulation in older adults. Amyloid beta protein is high in the brain of older adults with Alzheimer's disease. Hypertension may increase brain amyloid beta protein accumulation and affect memory and thinking ability in older adults. However, whether lowering blood pressure reduces brain amyloid beta protein and improves brain function is inconclusive.

The investigators hypothesize that treating high blood pressure alters brain pulsatility, which in turn reduces brain amyloid beta protein accumulation and improves brain structure and function.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55-79, all races/ethnicities, and both women and men are eligible;
2. Mini-mental state exam (MMSE) > 26 to exclude cognitive impairment or dementia;
3. Healthy normotensive subjects (24-hour ambulatory BP<125/75 mmHg without use of antihypertensive medication);
4. Patients with hypertension defined as 24-hour SBP ≥130 mmHg , patients on BP medications are eligible;
5. Patients with hypertension are willing to be randomized into either treatment group and ability to return to clinic or laboratory for follow-up visits over 12 months;
6. Fluency in English, adequate visual and auditory acuity to allow neuropsychological testing;
7. Screening laboratory tests and ECG without significant abnormalities that might interfere with the study

Exclusion Criteria:

1. History of stroke, transient ischemic attack, traumatic brain injury or severe cerebrovascular disease by clinical diagnosis or past MRI/CT;
2. Diagnosis of AD or other type of dementia and neurodegenerative diseases;
3. Evidence of severe depression or other DSM-V Axis I psychopathology
4. Unstable heart disease based on clinical judgment (heart attack/cardiac arrest, cardiac bypass procedures within previous 6 months and congestive heart failure), evidence of atrial fibrillation on ECG, or other severe medical conditions;
5. Chronic kidney diseases with GFR < 40 ml/min;
6. Orthostatic hypotension, defined as standing SBP<100 mmHg;
7. History of significant autoimmune disorders such as systemic lupus erythematosus, rheumatoid arthritis and polymyalgia rheumatica;
8. History of drug or alcohol abuse within the last 2 years;
9. Diagnosis of uncontrolled diabetes mellitus (fasting blood sugar ≥126 mg/dL or A1C >7.5%)
10. Obstructive sleep apnea;
11. Regularly smoking cigarette within the past year;
12. Severe obesity with BMI ≥ 45;
13. Participants enrolled in another investigational drug or device study within the past 2 months;
14. Carotid stent or sever stenosis (> 50%);
15. Pacemaker or other medical device of metal that precludes performing MRI;
16. History of B12 deficiency or hypothyroidism (stable treatment for at least 3 months is allowable);
17. Any conditions judged by the study investigators to be either medically inappropriate, or risky for participant or likely to have poor study adherence;
18. Claustrophobia;
19. Pregnancy

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rong Zhang, PhD, Principal Investigator — University of Texas Southwestern Medical Center and Texas Health Resources; Wanpen Vongpatanasin, MD, Principal Investigator — University of Texas Southwestern Medical Center; David Zhu, PhD, Principal Investigator — Michigan State University
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared approximately 18-24 months after the primary study publication.

REFERENCES:
- [Derived] Gottesman RF. To INFINITY and Beyond: What Have We Learned and What Is Still Unknown About Blood Pressure Lowering and Cognition? Circulation. 2019 Nov 12;140(20):1636-1638. doi: 10.1161/CIRCULATIONAHA.119.042827. Epub 2019 Nov 11. No abstract available. PMID 31710528

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 85 participants enrolled include 40 (Control group subjects-no intervention) and 45 participants (undergo intervention). These 45 subjects are randomized to either Standard care or Intensive care interventions that is summarized in the table below. Control group was not randomized and they did not receive an experimental intervention but received SOC.
Groups:
- Control Group: Control group subjects-no intervention- not randomized. This includes Healthy normotensive subjects (24-hour ambulatory BP<125/75 mmHg without use of antihypertensive medication) who undergo MRI as part of standard of care (SOC).
Period: Overall Study
Arm/Group | Standard Care | Intensive Treatment | Control Group
Started | 19 | 26 | 40
Completed | 17 | 22 | 40
Not Completed | 2 | 4 | 0

BASELINE CHARACTERISTICS:
Population: 85 participants enrolled include 40 (Control group subjects-no intervention) and 45 participants (undergo intervention). These 45 subjects are randomized to either Standard care or Intensive care interventions that is summarized in the table below. The baseline characteristics of the 40 subjects in Control group (no intervention) were not collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Intensive Treatment | Control Group | Total
Number analyzed (Participants) | 19 | 26 | 40 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 18 | 19 | 42
  >=65 years | 14 | 8 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (5.8) | 62.8 (6.4) | 60.3 (6.6) | 65.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 16 | 22 | 47
  Male | 10 | 10 | 18 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 2 | 11
  White | 12 | 21 | 35 | 68
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 26 | 40 | 45

OUTCOME MEASURES:

1. Primary Outcome: Changes in Gray Matter Intracranial Pulsatility
Description: Changes (12 month timepoint minus baseline) in intracranial pulsatility will be measured with CINE phase-contrast MRI. We will use the velocity-encoded CINE PC MRI to measure intracranial pulsatility. Pulsatility measured in mm per cardiac cycle
Time Frame: Baseline and 12-months
Population: Data was not collected for the Control group subjects since the investigator never planned to assess this outcome measure using Control group subject data as part of the pre-specified outcomes in the protocol.
Measure: Mean (Standard Deviation); unit: mm/cardiac cycle
Arm/Group | Standard Care | Intensive Treatment
Number analyzed (Participants) | 19 | 26
mm/cardiac cycle | -0.09 (0.04) | 0.02 (0.03)

2. Secondary Outcome: Changes in Overall Average 24 Hour Systolic Blood Pressure
Description: changes in overall average 24 hr ambulatory systolic blood pressure will be assessed SpaceLabs monitor
Time Frame: Baseline and 12-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Standard Care | Intensive Treatment
Number analyzed (Participants) | 19 | 26
mmHg | 17.9 (3.3) | 23.6 (2.8)

3. Secondary Outcome: Changes in Overall Average 24hr Diastolic Blood Pressure
Description: changes in overall average 24 hr ambulatory diastolic blood pressure will be assessed SpaceLabs monitor
Time Frame: Baseline and 12-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Standard Care | Intensive Treatment
Number analyzed (Participants) | 19 | 26
mmHg | 10.9 (1.5) | 12 (1.2)

4. Secondary Outcome: Regional Cortical Thickness Via Magnetic Resonance Imaging (MRI)
Time Frame: Baseline and 12-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Standard Care | Intensive Treatment | Control Group
Number analyzed (Participants) | 15 | 22 | 0
mm
  Baseline | 2.3 (0.09) | 2.4 (0.08) |
  12 month | 2.3 (0.09) | 2.3 (0.09) |

5. Secondary Outcome: Brain White Matter Hyperintensity (WMH) Via Magnetic Resonance Imaging (MRI)
Description: White matter hyperintensities (WMH) on brain T2 fluid-attenuated inversion recovery (FLAIR) magnetic resonance images (MRI) are commonly observed in older adults over 65 years old, and more extensive in those with vascular or Alzheimer's disease type of dementia. Qualitative and quantitative WMH characterization has been used as a biomarker to assist cerebral small vessel disease diagnosis and to assess treatment effects. In this report, the size of the WMH has been assessed with the PGS software, the top performer of the deep-learning algorithms from the 2017 MICCAI WMH segmentation challenge. The unit of the WMH total size presented in this report is in mL.
Time Frame: Baseline and 12-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Standard Care | Intensive Treatment | Control Group
Number analyzed (Participants) | 15 | 22 | 0
ml
  Baseline | 7.9 (12.9) | 2.8 (3.2) |
  12 Month | 7.5 (13.0) | 2.6 (2.9) |

6. Secondary Outcome: Brain White Matter Microstructural Integrity Via Magnetic Resonance Imaging (MRI)
Description: Fractional Anisotropy (FA) values are a measure of how directed diffusion is in a tissue, typically ranging from 0 to 1. A value of 0 indicates isotropic diffusion (diffusion is the same in all directions), while a value of 1 indicates highly anisotropic diffusion (diffusion is restricted to a single direction). FA is often used in diffusion tensor imaging (DTI) and is thought to reflect fiber density, axonal diameter, and myelination in white matter.
Time Frame: Baseline and 12-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Mean fractional anisotropy from DTI
Arm/Group | Standard Care | Intensive Treatment | Control Group
Number analyzed (Participants) | 15 | 22 | 0
Mean fractional anisotropy from DTI
  Baseline | 0.4 (0.02) | 0.4 (0.02) |
  12 Month | 0.4 (0.01) | 0.4 (0.01) |

7. Secondary Outcome: Brain Neural Network Functional Connectivity Via Magnetic Resonance Imaging (MRI)
Description: The brain's functional connectivity, particularly within the Default Mode Network (DMN), can be assessed using functional magnetic resonance imaging (fMRI) through the correlations between the activity of the brain regions within a network. In this report, the DMN regions were identified with a seed-based approach from another clinical trial with 420 subjects of a similar population. By identifying regions of interest (ROIs) within the DMN, researchers can analyze how these regions connect and interact with each other, revealing information about brain activity and potentially aiding in the diagnosis and understanding of various neurological and psychiatric conditions. Here, the functional connectivity of the DMN brain regions is reported in the unit of Pearson correlation R, with a range of 0 to 1 in this application. A high R value indicates a high level of connectivity.
Time Frame: Baseline and 12-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Pearson correlation R (r value)
Arm/Group | Standard Care | Intensive Treatment | Control Group
Number analyzed (Participants) | 14 | 21 | 0
Pearson correlation R (r value)
  Baseline | 0.39 (0.083) | 0.42 (0.14) |
  12 Month | 0.39 (0.079) | 0.4 (0.08) |

8. Secondary Outcome: NIH PROMIS Patient-reported Outcome Measures of Physical Health
Description: PROMIS® (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. Four items are used to assess global physical health. Three of these are administered using five-category response scales, and one item (rating of pain on average) uses a response scale of 0-10 that is recoded to five categories (0 = 1; 1-3 = 2; 4-6 = 3; 7-9 = 4; 10 = 5). T-score Metric: PROMIS measures use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. On the T-score metric:
  A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population. For PROMIS measures, higher scores equals more of the concept being measured (e.g., more Fatigue, more Physical Function).A score of 60 is one standard deviation above the average population
Time Frame: Baseline and 12-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Standard Care | Intensive Treatment | Control Group
Number analyzed (Participants) | 17 | 24 | 0
T score
  Baseline | 52.1 (6.4) | 51.0 (6.3) |
  12 Month | 50.9 (7.5) | 51.8 (7.4) |

9. Secondary Outcome: NIH PROMIS Patient-reported Outcome Measures of Mental Health
Description: PROMIS® (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. Four items are used to assess global physical health. Three of these are administered using five-category response scales, and one item (rating of pain on average) uses a response scale of 0-10 that is recoded to five categories (0 = 1; 1-3 = 2; 4-6 = 3; 7-9 = 4; 10 = 5). T-score Metric: PROMIS measures use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. On the T-score metric: A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population. For PROMIS measures, higher scores equals more of the concept being measured (e.g., more Fatigue, more Physical Function). A score of 60 is one standard deviation above the average population
Time Frame: Baseline and 12-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T sore
Arm/Group | Standard Care | Intensive Treatment | Control Group
Number analyzed (Participants) | 17 | 24 | 0
T sore
  Baseline | 56.0 (7.5) | 52.1 (7.4) |
  12 Month | 54.9 (8.4) | 54.0 (6.3) |

ADVERSE EVENTS:
Time Frame: 12 months
Description: Participants enrolled include Control group subjects (no intervention) and participants who underwent intervention. AEs monitored and collected for the subjects who were randomized to either Standard care or Intensive care interventions are summarized in the table below. The AEs for subjects in the Control group (no intervention) were not monitored and collected.
Arm/Group | Standard Care | Intensive Treatment
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/26
Other Adverse Events (participants affected / at risk) | 8/19 | 7/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=19) | Intensive Treatment (N=26)
Abnormal laboratory measure (General disorders) | 0 (0) | 1 (1) — low serum sodium
Orthostatic hypotension (General disorders) | 2 (2) | 1 (1)
Dizziness (General disorders) | 1 (1) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/43/NCT03354143/Prot_SAP_000.pdf